CLINICAL TRIAL: NCT02656901
Title: Incidence of Early Postoperative Cognitive Dysfunction After Closed Loop Anesthesia vs Inhalational Anesthesia or TIVA
Brief Title: Early Postoperative Cognitive Dysfunction After Closed Loop Anesthesia vs Inhalational Anesthesia or TIVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Foggia (Other)
Responsible Party: Principal Investigator, Cotoia Antonella, Prof., University of Foggia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 43/CE/2014
Record Dates: First submitted 2016-01-11; First posted 2016-01-15 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-05

CONDITIONS: Postoperative Cognitive Dysfunction
MeSH Terms: conditions — Postoperative Cognitive Complications

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (4):
- Auto Total endovenous anesthesia (Active Comparator): The closed loop delivering as already approved by ClinicalTrials.gov Identifier: NCT00392158
  Interventions: Device: auto total endovenous anesthesia
- Manual Desflurane anesthesia (Sham Comparator): The anesthesia will be maintained with desflurane to target the BIS of 50.
  Interventions: Device: Manual Desflurane anesthesia
- Manual sevoflurane anesthesia (Sham Comparator): The anesthesia will be maintained with sevoflurane to target the BIS of 50.
  Interventions: Device: Manual Sevoflurane anesthesia
- Manual total endovenous anestesia (Sham Comparator): In ManualTIVA group, the anesthesia will be maintained with propofol to target the BIS of 50
  Interventions: Device: Manual total endovenous anesthesia

INTERVENTIONS:
Device: auto total endovenous anesthesia — a closed-loop controller guided by the BIS steering the infusion pumps (Alaris Medical UK Ldt, Hants, Uk) as already approved by ClinicalTrials.gov Identifier: NCT00392158
  Other Names: AutoTIVA
  Arms: Auto Total endovenous anesthesia
Device: Manual Desflurane anesthesia — General anesthesia will be maintained with desflurane (Baxter D-Vapor Desflurane Vaporiser) to obtain a BIS value as close as possible to 50 and between 40
  Other Names: DES
  Arms: Manual Desflurane anesthesia
Device: Manual Sevoflurane anesthesia — General anesthesia will be maintained with sevoflurane ( Baxter Vapour 2000 Sevoflurane Vapouriser) to obtain a BIS value as close as possible to 50 and between 40 and 60.
  Other Names: SEVO
  Arms: Manual sevoflurane anesthesia
Device: Manual total endovenous anesthesia — In ManualTIVA group, the anesthesia will be maintained with propofol (Injectomat TIVA Agilia, Fresenius Kabi, Bad Hamburg, Germany) to obtain a BIS value as close as possible to 50 and between 40 and 60.
  Other Names: Manual TIVA
  Arms: Manual total endovenous anestesia

SUMMARY:
This study is designed to test the hypothesis that closed loop system reduces post operative cognitive dysfunction incidence 15 min after anesthesia more than desflurane, sevorane, total intravenous anesthesia manually guided by bispectral index in urologic surgical patients.

The secondary aim is to evaluate the postoperative cognitive impairment in in elderly vs younger surgical patients.

DETAILED DESCRIPTION:
Postoperative cognitive dysfunction (POCD) is a transient cognitive impairment manifested by compromised memory and concentration with altered performance on intellectual tasks that can affect patients of any age but it is more frequent in advanced age people after anesthesia.

Recently clinical research has demonstrated the efficacy of computer- controlled endovenous drug delivery system guided by bispectral index score (BIS) of the electroencephalogram as the control variable. The BIS closed loop (CL) titration of propofol and remifentanyl target control infusion provides clinically adequate anesthesia with stability of cardiovascular parameters and favorable patients outcomes, including decreasing drug consumption and shortened postoperative recovery times when compared with manual control infusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged above 18 years
* Patients undergoing elective urologic surgery under general anesthesia expected 2 hours
* American Society of Anesthesiology physical status II- III

Exclusion Criteria:

* Patients with body mass index greater than 30,
* Patients with clinically significant cardiopulmonary, hepatic, renal disorders, neurological, psychiatric or metabolic disease
* Patients unable to read and write and with impaired hearing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2016-01; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline of the Mini-Mental test examination score 15 min post anesthesia | 15 minutes before anesthetic procedures and 15 min after the end of general anesthesia
  The Mini-Mental State Examination (MMSE) test will be given 15 min before the anesthetic procedure and 15 min after the end of anesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Antonella Cotoia, MD, PhD, Principal Investigator — University of Foggia
Locations (1):
- University of Foggia, Foggia, Foggia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Liu N, Chazot T, Genty A, Landais A, Restoux A, McGee K, Laloe PA, Trillat B, Barvais L, Fischler M. Titration of propofol for anesthetic induction and maintenance guided by the bispectral index: closed-loop versus manual control: a prospective, randomized, multicenter study. Anesthesiology. 2006 Apr;104(4):686-95. doi: 10.1097/00000542-200604000-00012. PMID 16571963
- [Result] Liu N, Chazot T, Hamada S, Landais A, Boichut N, Dussaussoy C, Trillat B, Beydon L, Samain E, Sessler DI, Fischler M. Closed-loop coadministration of propofol and remifentanil guided by bispectral index: a randomized multicenter study. Anesth Analg. 2011 Mar;112(3):546-57. doi: 10.1213/ANE.0b013e318205680b. Epub 2011 Jan 13. PMID 21233500
- [Result] Liu N, Chazot T, Trillat B, Michel-Cherqui M, Marandon JY, Law-Koune JD, Rives B, Fischler M; Foch Lung Transplant Group. Closed-loop control of consciousness during lung transplantation: an observational study. J Cardiothorac Vasc Anesth. 2008 Aug;22(4):611-5. doi: 10.1053/j.jvca.2008.04.022. Epub 2008 Jun 25. PMID 18662642
- [Result] Liu N, Lory C, Assenzo V, Cocard V, Chazot T, Le Guen M, Sessler DI, Journois D, Fischler M. Feasibility of closed-loop co-administration of propofol and remifentanil guided by the bispectral index in obese patients: a prospective cohort comparison. Br J Anaesth. 2015 Apr;114(4):605-14. doi: 10.1093/bja/aeu401. Epub 2014 Dec 10. PMID 25500680